CLINICAL TRIAL: NCT04902768
Title: APPROACH-IS II: Assessment of Patterns of Patient Reported Outcomes in Adults With Congenital Heart Disease - International Study II
Brief Title: Assessment of Patterns of Patient Reported Outcomes in Adults With Congenital Heart Disease - International Study II
Acronym: APPROACH-IS II
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Philip Moons, Prof. Dr. Philip Moons, KU Leuven
Other Study IDs: S62537
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Quality of life; Patient reported outcomes; Patient reported experience measures; Geriatric phenotype
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with congenital heart disease
  Interventions: Other: This is an observational study, there is no intervention

INTERVENTIONS:
Other: This is an observational study, there is no intervention — This is an observational study, there is no intervention. Hence, this is not applicable.

SUMMARY:
This is an international, cross-sectional and descriptive study that aims to investigate differences in patient-reported outcome measures (PROMs) and patient-reported experience measures (PREMs) and that aims to explore the profile and healthcare needs of adults with congenital heart diseases.

DETAILED DESCRIPTION:
The research aims of this study are:

1. To further explore differences in a modified selection of patient-reported outcome measures (PROMs) and (as a new addition in APPROACH-IS II) explore differences in patient-reported experience measures (PREMs), by enrolling adults with congenital heart diseases in low, middle, and high income countries and including new potential explanatory variables ("Part 1").
2. To explore the profile and healthcare needs of a subgroup of older adults with congenital heart disease, with a particular focus on investigating the frailty phenotype ("Part 2").

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital heart disease, defined as: "a gross structural abnormality of the heart and/or intra-thoracic great vessels that is actually or potentially of functional significance (including mild, moderate, and complex heart defects)"
* Aged 18 years of age or older at the moment of study inclusion
* Diagnosed with congenital heart disease before the age of 10 years
* Follow-up at an ACHD center or included in a national/regional registry
* Physical, cognitive, and language abilities to complete self-report questionnaires

Exclusion Criteria:

- Prior heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with congenital heart disease who are in follow-up at an adult congenital heart disease center or included in a national/regional registry.
  For Part 1 of this study, each participating center will aim to recruit 200 adult patients with CHD aged 18 years or older with simple, moderate, or complex congenital heart disease. For Part 2 of this study, within these samples of 200 patients, centers will aim to recruit about 20 adults aged 40-50y, 20 adults aged 50-60y and 20 adults aged >60 years who are diagnosed with moderate to great disease complexity.
  Depending on the data collection method, sampling is at random or consecutive. Both a probability and convenience sample can be used.
Sampling Method: Probability Sample
Enrollment: 8415 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Patient-reported health status | Baseline
  This outcome is measured using the shortened version of the RAND-36. Composite physical (PCS) and mental health (MCS) scores are computed. Scores range from 0 (lowest health level) to 100 (highest health level).
Patient-reported health status | Baseline
  This outcome is measured using the Linear Analogue Scale Health Status (LAS HS). Scores range from 0 (worst imaginable health state) to 100 (best imaginable health state).
Patient-reported depressive symptoms | Baseline
  This outcomes is measured using the Patient Health Questionnaire 8. Scores range from 0 to 24. Scores of ≥10 indicate depression.
Patient-reported anxiety symptoms | Baseline
  This outcome is measured using the General Anxiety Disorder 7. Scores range from 0 to 21. Scores of 5, 10, and 15 are taken as cut-off points for mild, moderate and severe anxiety.
Patient-reported quality of life | Baseline
  This outcome is measured using the Linear Analog Scale on Quality of Life (LAS QOL). Scores range from 0 (worst imaginable quality of life) to 100 (best imaginable quality of life).
Patients' perception of providers' autonomy support | Baseline
  This outcome is measured using the modified Health Care Climate Questionnaire (mHCCQ). Each of the 6 items is scored from 1 to 7. Scores are calculated by averaging the individual item scores. Higher average score represents a higher level of perceived autonomy support.
Cognitive functioning | Baseline
  This outcome is measured using the Montreal Cognitive Assessment Screener (MoCA). Scores range from 0 to 30. Scores of <26 indicate cognitive dysfunction.
Frailty phenotype | Baseline
  This outcome is classified using the Fried method (i.e., non-frail (no positive criterion), pre-frail (1 or 2 criteria positive), or frail (when ≥3 criteria are positive).

SECONDARY OUTCOMES:
Patient-reported stigma | Baseline
  This outcome is measured using the Chronic Illness Stigma Scale (CISS). Scores range from 8 to 40. Higher scores indicating higher levels of perceived stigma.
Patient-reported illness identity | Baseline
  This outcome is measured using the Illness Identity Questionnaire (IIQ). The questionnaire consists of a five-item rejection scale, seven-item enrichment scale, five-item acceptance scale and eight-item engulfment scale. A mean score is calculated per subscale. Higher scores indicate more rejection, enrichment, acceptance or engulfment.
Patient-reported empowerment | Baseline
  This outcome is measured using the Gothenburg Empowerment Scale (GES generic v1.1). Scores range from 15 to 75. Higher score reflects a higher level of empowerment.
Patient-reported healthcare utilization | Baseline
  This outcomes was measured using the Patient-Reported Inpatient and outpatient Utilization Survey (PRIUS). Higher numbers indicate more healthcare use.
Patient-reported functional status | Baseline
  This outcome is classified according to the New York Heart Association (NYHA).
Patient-reported social support | Baseline
  This outcomes is measured using the Multidimensional Scale on Perceived Social Support Scale (MSPSS). Scores range from 12 to 84. Higher score indicates greater social support perceived by an individual.
Patient-reported parental involvement | Baseline
  This outcome is measured using an adapted version of the subscale on parents of the Multidimensional Scale on Perceived Social Support. Scores range from 5 to 35. Higher score indicates greater parental support in childhood and adolescence.
Advance care planning | Baseline
  This outcome is measured using a survey developed for APPROACH-IS II by the Steering Committee, based on previous research. A sample question is 'Have you personally written down information about the care you would want in case you become seriously ill in the future?'.
Patient-reported social media to connect with peers | Baseline
  This outcome is measured using a survey developed for APPROACH-IS II by the Steering Committee, based on previous research. A sample question is 'How would you describe your experiences connecting with other people with CHD through social media?'.
Presence and burden of comorbidities | Baseline
  This outcome is measured using the Charlson Comorbidity Index.
Patient-reported socio-demographic variables (eg. age, educational level) | Baseline
  Self-reported
Medical variables by chart review (eg. diagnosis, cardiac surgeries) | Baseline
  This outcome is classified according to the adult congenital heart disease anatomic and physiological (ACHD AP) classification system of Stout and colleagues.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Moons, PhD, RN, Principal Investigator — Professor in Healthcare Sciences
Locations (53):
- United States (10):
  - University of California, San Francisco, California
  - Lucile Packard Children's Hospital and Stanford Health Care, Stanford, California
  - University of Florida Health, Gainesville, Florida
  - Taussig Heart Center of Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's / Brigham and Women's, Boston, Massachusetts
  - Mount Sinai Heart, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Philadelphia Penn Medicine, Philadelphia, Pennsylvania
  - University of Southwestern Medical Center, Dallas, Texas
- Argentina (2):
  - Hospital San Juan De Dios De La Plata, Buenos Aires
  - Hospital de Niños, Córdoba
- Melbourne Children's Cardiology, Melbourne, Australia
- Vienna General Hospital, Vienna, Austria
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
- Princess Marina Hospital, Gaborone, Botswana
- Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto, Ribeirão Preto, Brazil
- National Heart Hospital, Sofia, Bulgaria
- Clinique Medical Le Jourdain, Yaoundé, Cameroon
- Canada (2):
  - Mazankowski Alberta Heart Institute, Edmonton
  - Montreal Heart Institute, Université de Montréal, Montreal
- Intituto Nacional Del Torax, Santiago, Chile
- Meintegral Clinic, Manizales, Colombia
- Copenhagen University Hospital, Copenhagen, Denmark
- College of Health sciences, Addis Ababa University, Addis Ababa, Ethiopia
- France (3):
  - Hôpital cardiologique Haut-Leveque, Bordeaux
  - Montpellier University Hospital, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
- AHEPA University Hospital, Thessaloniki, Greece
- Amrita Institute of Medical Sciences, Kochi, India
- Policlinico San Donato (IRCCS), Milan, Italy
- Chiba Cerebral and Cardiovascular Center, Chiba, Japan
- Paediatric & Congenital Heart Centre, IJN (National Heart Institute), Kuala Lumpur, Malaysia
- Mater Dei Hospital, Msida, Malta
- Centrum voor Congenital Hartafwijkingen, Groningen, Netherlands
- Oslo University Hospital, Rikshospitalet, Oslo, Norway
- Aga Khan University Hospital, Karachi, Pakistan
- Reference Center of Congenital Heart Disease , University Hospital Center of São João, Porto, Portugal
- Centre Hospitalier Régional de Thiès, Thiès, Senegal
- Samsung Medical Center, Seoul, South Korea
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Stockholm
  - Umea University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- Switzerland (3):
  - University Hospital Bern, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier universitaire vaudois, Lausanne
- National Taiwan University Hospital, Taipei, Taiwan
- Ege University Health Application and Research Center, Cardiology Department, Bornova, Turkey (Türkiye)
- United Kingdom (2):
  - Royal Brompton Hospital, Royal Brompton & Harefield Hospitals, Guy's and St Thomas' NHS Foundation Trust, London
  - Freeman Hospital, Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No
Well-argued and reasonable requests can be directed to the Principal Investigator (Prof. Philip Moons) of the study.

REFERENCES:
- [Derived] van Bulck L, Goossens E, Kovacs AH, Luyckx K, Ladak LA, Leye M, van de Bruaene A, Leong MC, Kaneva A, Pavao RB, Araujo JJ, Sasikumar N, Gabriel H, Goshu DY, Lu CW, Enomoto J, Areias ME, Kosmidis D, Coats L, Valente AM, Moon JR, Ladouceur M, Thomet C, Jackson JL, Sandberg C, Callus E, Kim YY, Lykkeberg B, Alday L, Bredy C, Saidi A, Reyes FB, Menahem S, de Hosson M, Mandelenakis Z, Christersson C, Zaidi A, Johansson B, Andresen B, Ambassa JC, Mattsson E, Constantine A, Amedro P, van Melle JP, Cedars A, Ortiz L, Demir F, Khairy P, Windram J, Bouchardy J, Caruana M, Jameson SM, Mahadevan VS, McGrath LB, Mwita JC, Moons P; APPROACH-IS II consortium, International Society for Adults Congenital Heart Disease (ISACHD). Advance Care Planning in Adults With Congenital Heart Diseases: Current Practices, Preferences, and Needs of 8,281 Adults From 32 Countries. Can J Cardiol. 2026 Jan 8:S0828-282X(25)01607-1. doi: 10.1016/j.cjca.2025.12.039. Online ahead of print. PMID 41519299
- [Derived] Ansari Ramandi MM, Van Bulck L, Ceelen DCH, Voors AA, Goossens E, Kovacs AH, Luyckx K, Van De Bruaene A, Gabriel H, Lykkeberg B, Thomet C, de Hosson M, Ladouceur M, Saidi A, Kosmidis D, Areias ME, Miranda J, Sandberg C, Mandalenakis Z, Coats L, Amedro P, Khairy P, Valente AM, Johansson B, Kaneva A, Andresen B, Christersson C, Baraona Reyes F, Hlebowicz J, Enomoto J, Kim YY, Menahem S, Yang HL, Moon JR, Bredy C, Schmidt A, Callus E, Araujo JJ, Constantine A, Zaidi A, Bouchardy J, Jameson SM, Kutty S, McGrath LB, Leong MC, Ortiz L, Demir Korkmaz F, Caruana M, Leye M, Moons P, van Melle JP; APPROACH-IS II Consortium; International Society for Adults With Congenital Heart Disease. Quality of Life in Adults With Transposition of the Great Arteries With a Systemic Right or Left Ventricle. Can J Cardiol. 2025 Dec;41(12):2544-2553. doi: 10.1016/j.cjca.2025.09.010. Epub 2025 Sep 15. PMID 40962221
- [Derived] Moons P, Kovacs AH, Goossens E, Luyckx K, Ladak L, Leye M, Van De Bruaene A, Leong MC, Kaneva A, Manso PH, Araujo JJ, Sasikumar N, Gabriel H, Yadeta D, Wang JK, Enomoto J, Areias ME, Kosmidis D, Coats L, Valente AM, Moon JR, Ladouceur M, Thomet C, Jackson JL, Sandberg C, Callus E, Kim YY, Lykkeberg B, Alday L, Bredy C, Saidi A, Baraona Reyes F, Menahem S, de Hosson M, Hlebowicz J, Christersson C, Zaidi AN, Johansson B, Andresen B, Ambassa JC, Mattsson E, Constantine A, Amedro P, van Melle JP, Kutty S, Ortiz L, Demir F, Khairy P, Windram J, Bouchardy J, Caruana M, Jameson SM, Mahadevan VS, McGrath LB, Mwita JC, Van Bulck L; APPROACH-IS II consortium, on behalf of the International Society for Adults Congenital Heart Disease (ISACHD). Perceived health, psychological distress and quality of life in 8415 adults with congenital heart disease from 32 countries. Heart. 2025 Aug 12;111(17):818-827. doi: 10.1136/heartjnl-2024-325296. PMID 40579213
- [Derived] Moons P, Goossens E, Luyckx K, Kovacs AH, Andresen B, Moon JR, Van De Bruaene A, Rassart J, Van Bulck L; APPROACH-IS II consortium and ISACHD. The COVID-19 pandemic as experienced by adults with congenital heart disease from Belgium, Norway, and South Korea: impact on life domains, patient-reported outcomes, and experiences with care. Eur J Cardiovasc Nurs. 2022 Aug 29;21(6):620-629. doi: 10.1093/eurjcn/zvab120. PMID 34927192